CLINICAL TRIAL: NCT07179601
Title: Hemorrhoidal Artery Embolization: Longitudinal Impact On Symptoms (HELIOS)
Acronym: HELIOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Lucas R. Cusumano, MD, Interventional Radiologist, Assistant Clinical Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-0704
Record Dates: First submitted 2025-09-16; First posted 2025-09-18 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-10

CONDITIONS: Internal Hemorrhoids; HAE

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Hemorrhoidal artery embolization (Experimental): Patients in this arm will undergo hemorrhoidal artery embolization (HAE) for treatment of symptomatic internal hemorrhoids
  Interventions: Procedure: Hemorrhoidal artery embolization

INTERVENTIONS:
Procedure: Hemorrhoidal artery embolization — Hemorrhoidal artery embolization (HAE) involves the deliberate blockage of enlarged rectal or hemorrhoidal arteries leading to reduction of abnormal blood flow to the hemorrhoidal tissue. The aim of HAE is to the improve symptoms related to internal hemorrhoids, especially bleeding.

SUMMARY:
Hemorrhoidal artery embolization (HAE) is a novel treatment for symptomatic internal hemorrhoids. HAE involves the deliberate blockage (embolization) of enlarged rectal or hemorrhoidal arteries leading to reduction of abnormal blood flow to the hemorrhoidal tissue. The aim of HAE is to the improve hemorrhoid related symptoms, especially bleeding. Initial reports of HAE have demonstrated that it both safe and effective. Following an initial clinic visit to determine trial candidacy, enrolled patients will be subsequently treated with HAE. Patients will be followed for a year with clinic follow-up visits at 1, 3, 6 and 12 months.

DETAILED DESCRIPTION:
Hemorrhoidal artery embolization (HAE) is a novel treatment for symptomatic internal hemorrhoids. HAE involves the deliberate blockage (embolization) of enlarged rectal or hemorrhoidal arteries leading to reduction of abnormal blood flow to the hemorrhoidal tissue. The aim of HAE is to the improve hemorrhoid related symptoms, especially bleeding. Initial reports of HAE have demonstrated that it both safe and effective. However, the initial data is limited due to variations in embolization techniques, few studies with prospective long-term follow-up, and studies focusing on patients with only severe symptoms. Further research is needed to understand the specific long-term effectiveness of different embolization materials in a population that more accurately reflects the large number of patients with hemorrhoidal disease who would likely benefit from HAE. The proposed research project includes 22 patients with symptomatic internal hemorrhoids. Following an initial clinic visit to determine trial candidacy, enrolled patients will be subsequently treated with HAE. Patients will be followed for a year with clinic follow-up visits at 1, 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 90 years
* Ability to give written informed consent and to comply with the follow-up visits
* Symptomatic hemorrhoidal disease with French Bleeding Score (FBS) of at least four out of nine
* Refusal of or contraindication to surgery
* Refusal of or contraindication to other minimally invasive hemorrhoid treatments
* Grade I to III hemorrhoids
* Previous anoscopy or colonoscopy demonstrating internal hemorrhoids within 1 year
* Supply of the CCR from either the SRA or MRA on intra-procedural angiogram prior to embolization

Exclusion Criteria:

* Asymptomatic patients
* Patients who ever had previous colorectal surgery
* Grade IV hemorrhoids
* Colorectal disease other than hemorrhoids that could result in bleeding
* Anatomic findings on CTA that would preclude successful embolization
* Contraindication to iodinated contrast
* Inability to give written informed consent
* Active infection or malignancy
* Recent (within 12 months) or active cigarette use
* History of inflammatory bowel disease
* Uncorrectable bleeding diathesis
* Presence of portal hypertension or rectal varices seen on pre-procedure CTA or anoscopy/colonoscopy
* No SRA or MRA supply to the CCR seen intra-procedural angiogram

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with decrease in bleeding related symptoms of internal hemorrhoids as defined as a two-point decrease in French Bleeding Score | From baseline to 12 months post procedure

SECONDARY OUTCOMES:
Proportion of technically successful HAE procedures | From baseline to 12 months post procedure
Change in non-bleeding related symptoms of internal hemorrhoids as measured by the Hemorrhoid Disease Symptom Score (HDSS) | From baseline to 12 months post procedure
  The Hemorrhoidal Disease Symptom Score (HHDS) is a widely used questionnaire used by health professionals to evaluate the condition of patients with hemorrhoids. It can be self-administered and asks patients to rate the frequency and intensity of five primary symptoms: pain, itching, bleeding, soiling, and prolapse. Each symptom is rated on a scale of 0 to 4, with 0 indicating no symptoms and 4 indicating the most severe symptoms. The total HDSS score ranges from 0 to 20, with higher scores indicating more severe hemorrhoidal disease.
Change in non-bleeding related symptoms of internal hemorrhoids as measured by the Short Health Scale-Hemorrhoidal Disease (SHSHD) | From baseline to 12 months post procedure
  The Short Health Scale-Hemorrhoidal Disease questionnaire is a validated tool used to assess the impact of hemorrhoidal disease on a patient's health-related quality of life. It can be self-administered and measures four key dimensions: symptom load, functional status, disease-specific worries, and general well-being. Each symptom is rated on a scale of 1 to 7, with 1 indicating no symptoms and 7 indicating the most severe symptoms. The total SHSHD score ranges from 4 to 28, with higher scores indicating more severe hemorrhoidal disease.
Change in pain related to as measured by the Visual Analog Scale (VAS) | From baseline to 12 months post procedure
  The Visual Analog Scale (VAS) is a validated commonly used pain score. The VAS ranges from 0 to 10, with higher scores indicated higher pain levels.
Change in concomitant hemorrhoid medical therapy | From baseline to 12 months post procedure
Level of patient satisfaction after HAE as determined by patient satisfaction questionnaire | From baseline to 12 months post procedure
  Patient satisfaction will be determined by a patient satisfaction questionnaire with the following four options: very satisfied, satisfied, a little satisfied, and unsatisfied
Proportion of patients requiring subsequent non-surgical internal hemorrhoid procedures | From baseline to 12 months post procedure
Proportion of patients requiring surgical management of their internal hemorrhoids | From baseline to 12 months post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Lucas Cusumano, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ganz RA. The evaluation and treatment of hemorrhoids: a guide for the gastroenterologist. Clin Gastroenterol Hepatol. 2013 Jun;11(6):593-603. doi: 10.1016/j.cgh.2012.12.020. Epub 2013 Jan 16. No abstract available. PMID 23333220
- [Background] Margetis N. Pathophysiology of internal hemorrhoids. Ann Gastroenterol. 2019 May-Jun;32(3):264-272. doi: 10.20524/aog.2019.0355. Epub 2019 Jan 23. PMID 31040623
- [Background] Hawkins AT, Davis BR, Bhama AR, Fang SH, Dawes AJ, Feingold DL, Lightner AL, Paquette IM; Clinical Practice Guidelines Committee of the American Society of Colon and Rectal Surgeons. The American Society of Colon and Rectal Surgeons Clinical Practice Guidelines for the Management of Hemorrhoids. Dis Colon Rectum. 2024 May 1;67(5):614-623. doi: 10.1097/DCR.0000000000003276. Epub 2024 Jan 31. No abstract available. PMID 38294832
- [Background] Cengiz TB, Gorgun E. Hemorrhoids: A range of treatments. Cleve Clin J Med. 2019 Sep;86(9):612-620. doi: 10.3949/ccjm.86a.18079. PMID 31498764
- [Background] Wald A, Bharucha AE, Cosman BC, Whitehead WE. ACG clinical guideline: management of benign anorectal disorders. Am J Gastroenterol. 2014 Aug;109(8):1141-57; (Quiz) 1058. doi: 10.1038/ajg.2014.190. Epub 2014 Jul 15. PMID 25022811
- [Background] Makris GC, Thulasidasan N, Malietzis G, Kontovounisios C, Saibudeen A, Uberoi R, Diamantopoulos A, Sapoval M, Vidal V. Catheter-Directed Hemorrhoidal Dearterialization Technique for the Management of Hemorrhoids: A Meta-Analysis of the Clinical Evidence. J Vasc Interv Radiol. 2021 Aug;32(8):1119-1127. doi: 10.1016/j.jvir.2021.03.548. Epub 2021 May 7. PMID 33971251
- [Background] Vidal V, Louis G, Bartoli JM, Sielezneff I. Embolization of the hemorrhoidal arteries (the emborrhoid technique): a new concept and challenge for interventional radiology. Diagn Interv Imaging. 2014 Mar;95(3):307-15. doi: 10.1016/j.diii.2014.01.016. Epub 2014 Feb 28. PMID 24589187
- [Background] Panneau J, Mege D, Di Bisceglie M, Duclos J, Habert P, Bartoli A, Vidal V, Tradi F. Rectal Artery Embolization for Hemorrhoidal Disease: Anatomy, Evaluation, and Treatment Techniques. Radiographics. 2022 Oct;42(6):1829-1844. doi: 10.1148/rg.220014. PMID 36190848
- [Background] Kucukay MB, Kucukay F. Superior Rectal Artery Embolization with Tris-Acryl Gelatin Microspheres: A Randomized Comparison of Particle Size. J Vasc Interv Radiol. 2021 Jun;32(6):819-825. doi: 10.1016/j.jvir.2021.02.011. Epub 2021 Feb 25. PMID 33640516
- [Background] Bagla S, Pavidapha A, Lerner J, Kasimcan MO, Piechowiak R, Josovitz K, Marathe A, Isaacson A, Sajan A. Outcomes of Hemorrhoidal Artery Embolization from a Multidisciplinary Outpatient Interventional Center. J Vasc Interv Radiol. 2023 May;34(5):745-749. doi: 10.1016/j.jvir.2023.01.023. Epub 2023 Feb 1. PMID 36736822
- [Background] Moussa N, Sielezneff I, Sapoval M, Tradi F, Del Giudice C, Fathallah N, Pellerin O, Amouyal G, Pereira H, de Parades V, Vidal V. Embolization of the superior rectal arteries for chronic bleeding due to haemorrhoidal disease. Colorectal Dis. 2017 Feb;19(2):194-199. doi: 10.1111/codi.13430. PMID 27338153
- [Background] Tradi F, Louis G, Giorgi R, Mege D, Bartoli JM, Sielezneff I, Vidal V. Embolization of the Superior Rectal Arteries for Hemorrhoidal Disease: Prospective Results in 25 Patients. J Vasc Interv Radiol. 2018 Jun;29(6):884-892.e1. doi: 10.1016/j.jvir.2018.01.778. Epub 2018 Apr 30. PMID 29724519
- [Background] Nguyenhuy M, Xu Y, Kok HK, Maingard J, Joglekar S, Jhamb A, Brooks M, Asadi H. Clinical Outcomes Following Rectal Artery Embolisation for the Treatment of Internal Haemorrhoids: A Systematic Review and Meta-Analysis. Cardiovasc Intervent Radiol. 2022 Sep;45(9):1351-1361. doi: 10.1007/s00270-022-03154-7. Epub 2022 May 12. PMID 35551442
- [Background] Moussa N, Bonnet B, Pereira H, Pechmajou L, Pellerin O, Abed A, Del Giudice C, Dean C, Bouda D, de Parades V, Fathallah N, Sapoval M. Mid-Term Results of Superior Rectal Artery and Coils for Hemorrhoidal Embolization with Particles Bleeding. Cardiovasc Intervent Radiol. 2020 Jul;43(7):1062-1069. doi: 10.1007/s00270-020-02441-5. Epub 2020 Apr 27. PMID 32342155